201330 [DTPA (BOOSTRIX)-048 PRI]
Statistical Analysis Plan Final

| | Statistical Analysis Plan Final |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A phase IV, open-label, non-randomised, multicentre study to assess the immunogenicity and safety of <i>Infanrix hexa</i> <sup>TM</sup> administered as primary vaccination in healthy infants born to mothers vaccinated with <i>Boostrix</i> <sup>TM</sup> during pregnancy or immediately postdelivery. |
| eTrack study number and<br>Abbreviated Title | 201330 [DTPA (BOOSTRIX)-048 PRI] |
| Scope: | All analyses as planned per protocol and for study report |
| Date of Statistical Analysis<br>Plan | 16-Jul-2018 Final |
| Co-ordinating author: | PPD |
| Reviewed by: | R&D Project Leader) PPD Lead (CRDL) PPD (Lead Statistician) PPD (Scientific writer) PPD (Regulatory Affair) PPD (Safety Scientist) VxRD Medical Vx Office of Medical Governance and Bioethics Public Disclosure Global (Public disclosure) |
| Approved by: | PPD (Clinical and Epidemiology R&D Project Leader) PPD , Clinical Research and Development Lead (CRDL) PPD (Scientific writer) PPD (Lead Statistical analyst) PPD (Lead Statistician) |
| APP 9000058193 | Statistical Analysis Plan Template (Effective date: 14 April 2017) |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | TIONS | 8 |
| 1. | DOC | JMENT HI | STORY | 10 |
| 2. | STUD | Y DESIGN | N | 10 |
| 3. | | CTIVES | | 1.1 |
| J. | 3.1. | | objective | |
| | 3.2. | • | ary objectives | |
| 4. | ENDF | OINTS | | 15 |
| | 4.1. | Primary of | endpoints | 15 |
| | 4.2. | Seconda | ary endpoints | 15 |
| 5. | | | S | |
| | 5.1. | | n | |
| | | 5.1.1. | All enrolled subjects | |
| | | 5.1.2.<br>5.1.3. | Total vaccinated cohort (TVC) | |
| | | 5.1.3.<br>5.1.4. | ATP cohort for analysis of safetyATP cohort for analysis of immunogenicity | |
| | 5.2. | - | for eliminating data from Analysis Sets | |
| | 0.2. | 5.2.1. | Elimination from Total vaccinated cohort (TVC) | |
| | | 5.2.2. | Elimination from ATP cohort for safety | |
| | | - | 5.2.2.1. Excluded subjects | |
| | | 5.2.3. | Elimination from ATP cohort for immunogenicity | |
| | | | 5.2.3.1. Excluded subjects | 18 |
| 6. | STAT | | NALYSES | |
| | 6.1. | | aphy | 20 |
| | | 6.1.1. | Analysis of demographics/baseline characteristics planned in the protocol | 20 |
| | | 6.1.2. | Additional considerations | |
| | 6.2. | - | e | |
| | 0.2. | 6.2.1. | Analysis of exposure planned in the protocol | |
| | | 6.2.2. | Additional considerations | |
| | 6.3. | Immunog | genicity | |
| | | 6.3.1. | Analysis of immunogenicity planned in the protocol | 21 |
| | | 6.3.2. | Additional considerations | |
| | 6.4. | • | of safety | 23 |
| | | 6.4.1. | Analysis of safety and reactogenicity planned in the protocol | 23 |
| | | 6.4.2. | Additional considerations | |
| | | 0.4.2. | 6.4.2.1. Combined Solicited and Unsolicited Adverse | |
| | | | Events | |
| 7. | ANAL | YSIS INTE | ERPRETATION | 25 |
| 8. | CONF | OUCT OF A | ANALYSES | 25 |
| | | | ce of analyses | |

| | | | CONFIDENTIAL | |
|---|---|---|---|---|
| | | | 201330 [DTPA (BOOSTRI)<br>Statistical Analysis | |
| | 8.2. | Statistic | al considerations for interim analyses | |
| 9. | CHAN | GES FRO | OM PLANNED ANALYSES | 26 |
| 10. | LIST | OF FINAL | REPORT TABLES, LISTINGS AND FIGURES | 28 |
| 11. | | | NDARD DATA DERIVATION RULE AND STATISTICAL | |
| | METH | IODS | | 29 |
| | 11.1. | Statistic | al Method References | 29 |
| | 11.2. | Standar | d data derivation | 29 |
| | | 11.2.1. | Date derivation | 29 |
| | | 11.2.2. | Dose number | 29 |
| | | 11.2.3. | Demography | 30 |
| | | 11.2.4. | | |
| | | 11.2.5. | | |
| | | 11.2.6. | • | |
| 12 | ∧ NINI⊏ | V 2: CTII | DV SDECIEIC MOCK TEI | 35 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## **LIST OF TABLES**

| | | PAGE |
|---|---|---|
| Table 1 | Study groups and epoch foreseen in the study | 12 |
| Table 2 | Study groups and treatments foreseen in the study | 12 |
| Table 3 | Blinding of study epoch | 12 |
| Table 4 | Intensity scales for solicited symptoms in infants less than 6 years of age | 33 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design diagram for infants receiving a 3-dose schedule of Infanrix hexa | 10 |
| igure 2 | Study design diagram for infants receiving a 2-dose schedule of<br>Infanrix hexa | 11 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## **LIST OF TEMPLATES**

| | Ρ. | AGE |
|---|---|---|
| Template 1 | Number of subjects enrolled by center (Total vaccinated cohort) | 35 |
| Template 2 | Number of subjects enrolled by country (Total vaccinated cohort) | 36 |
| Template 3 | Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Total vaccinated cohort) | 36 |
| Template 4 | Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort) | 37 |
| Template 5 | Number of subjects enrolled into the study as well as excluded from ATP analyses with reasons for exclusion | 38 |
| Template 6 | Deviations from specifications for age and intervals between study visits for subjects vaccinated with Infanrix hexa(<2> dose schedule - 1 dose/visit) (Total Vaccinated Cohort) | 39 |
| Template 7 | Summary of demographic characteristics (Total vaccinated cohort) | 40 |
| Template 8 | Summary of vital signs characteristics (Total Vaccinated Cohort) | 41 |
| Template 9 | Study population (TVC) | 42 |
| Template 10 | Seropositivity rates and GMCs for anti-PT, anti-FHA and anti-PRN antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity) | 42 |
| Template 11 | Seropositivity, seroprotection and GMC rates for <anti-tetanus> antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity)</anti-tetanus> | 43 |
| Template 12 | Seroprotection rates for anti-poliovirus type 1,2,3 antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity) | 44 |
| Template 13 | Vaccine responses for anti-PT, anti-FHA and anti-PRN antibody concentration 1 month after the last dose of the primary vaccination course (ATP cohort for immunogenicity) | 45 |
| Template 14 | Reverse cumulative curve for anti-diphtheria antibody concentration before first dose and 1 month post last dose of the primary vaccination course (ATP cohort for immunogenicity) | 46 |
| Template 15 | Number and percentage of subjects who received study vaccine doses by vaccination group (Total vaccinated cohort) | 47 |
| Template 16 | Compliance in returning symptom sheets (Total vaccinated cohort) | 47 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

| Template 17 | Percentage and nature of <grade 3="">symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort)</grade> | 48 |
|---|---|---|
| Template 18 | Percentage of solicited local symptoms reported during the 4-day (Day 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort) | 49 |
| Template 19 | Percentage of solicited general symptoms reported during the 4-day (Days 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort) | 52 |
| Template 20 | Percentage of Unsolicited symptoms experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) after any dose (Total vaccinated cohort). | 54 |
| Template 21 | Number (%) of subjects with serious adverse events from the Day 0 to end of the study (Total Vaccinated cohort) | 54 |
| Template 22 | Solicited and unsolicited adverse events experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort) | 55 |
| Template 23 | Number and percentage of subjects taking a concomitant medication and antipyretic medication during the 4-day (Days 0-3) follow-up period post-vaccination by dose and overall (Total vaccinated cohort) | 56 |
| Template 24 | Minimum and maximum activity dates (Total vaccinated cohort) | 56 |
| Template 25 | Number of enrolled subjects by age category at visit1 | 57 |
| Template 26 | Listing of SAEs from Day 0 up study (Total vaccinated cohort) | 57 |
| Template 27 | Listing of dropouts due to AEs, SAEs and solicited symptoms (Total vaccinated cohort) | 57 |

## 201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

#### **LIST OF ABBREVIATIONS**

AE Adverse event

Anti-HBs Antibodies against hepatitis B surface antigen

ATP According-To-Protocol

CI Confidence Interval

CRDL Clinical Research and Development Lead

CRF Case Report Form

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

dTpa Combined reduced antigen content diphtheria-tetanus-acellular

pertussis vaccine

DTPa Diphtheria-Tetanus-acellular Pertussis

eCRF electronic Case Report Form

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

EOS End of study

EPAR European Public Assessment Report

FHA Filamentous Haemagglutinin

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

HBs Hepatitis B surface antigen

HBV Hepatitis B Virus

Hib Haemophilus influenzae type b

IDMC Independent Data Monitoring Committee

IM Intramuscular

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

IMP Investigational Medicinal Product

IPV Inactivated Poliovirus Vaccine

IU/ml International units per milliliter

LAR Legally Acceptable Representative

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable

PRN Pertactin

PRP Hib capsular polysaccharide Polyribosyl-Ribitol Phosphate

PT Pertussis Toxoid

SAE Serious adverse event

SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

SRT Safety Review Team

TFL Tables Figures and Listings

TOC Table of Content

TVC Total Vaccinated Cohort

UL Upper Limit of the confidence interval

WHO World Health Organization

#### 1. DOCUMENT HISTORY

| Date Description Protocol Version | | Protocol Version |
|---|---|---|
| 16-JUL-2018 | Final Version | Amendment 1 Final - 06-SEP-2016 |

## 2. STUDY DESIGN

Figure 1 Study design diagram for infants receiving a 3-dose schedule of Infanrix hexa



N: Maximum number of subjects planned to be enrolled

M = Month, Mo = age in months

Timepoints have been numbered based on the different vaccination schedules. D0, M1, M2 and M3 timepoints reflect for subjects who will be vaccinated according to the 2, 3 and 4 month schedule while D0, M2, M4 and M5 timepoints reflect for subjects who will be vaccinated according to the 2, 4 and 6 month schedule.

\* In some countries/regions with an *Infanrix hexa* 3-dose schedule, *Prevenar* 13 is given as a 2-dose schedule at 2 and 4 months of age as a part of the routine immunisation programme

Pre-Pri = Blood sample to be collected before the first dose of the primary vaccination course

Post-Pri = Blood sample to be collected one month after the last dose of the primary vaccination course

Figure 2 Study design diagram for infants receiving a 2-dose schedule of Infanrix hexa



N: Maximum number of subjects planned to be enrolled

M = Month, Mo = age in months

Pre-Pri = Blood sample to be collected before the first dose of the primary vaccination course
Post-Pri = Blood sample to be collected one month after the last dose of the primary vaccination course
Subjects will be vaccinated either at 2 and 4 months of age or 3 and 5 months of age, according to the routine national immunisation schedule

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of the protocol), are essential and required for study conduct.

- Experimental design: Phase IV, open-label, non-randomised, multi-centric, multi-country study with two parallel groups.
- Duration of the study: The intended duration of the study is approximately 3 months, per subject, for subjects vaccinated according to the 2 and 4, the 3 and 5 or the 2, 3 and 4 months schedule and approximately 5 months, per subject, for those vaccinated according to 2, 4 and 6 month schedule.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

- Epoch 001: Primary starting at Visit 1 (Day 0) and ending at Visit 4 (Month 3 or 5, depending on the vaccination schedule).
- End of study (EOS): Last testing results released of samples collected at Visit 4.
- Study groups: The study groups and epoch foreseen in the study are presented in Table 1.

Table 1 Study groups and epoch foreseen in the study

| Study Groups | Number of subjects | Age (Min - Max)* | Epoch Epoch 001 |
|---------------|--------------------|--------------------|-----------------|
| dTpa Group | 340 | 6- <b>14</b> weeks | X |
| Control Group | 340 | 6- <b>14</b> weeks | X |

<sup>\*</sup>Up to and including 14 weeks and 6 days of age.

The study groups and treatment foreseen in the study are presented in Table 2.

Table 2 Study groups and treatments foreseen in the study

| Treetment names | Vaccine name | Study Groups | |
|-----------------|-----------------------|--------------|---------------|
| Treatment names | vaccine name | dTpa Group | Control Group |
| Infanrix hexa | DTP <b>a</b> -HBV-IPV | Х | X |
| | Hib | Х | X |
| Prevenar 13 | Prevenar 13 | Х | X |

- Control: uncontrolled
- Vaccination schedules: All subjects will receive either 3 doses of *Infanrix hexa* coadministered with *Prevenar* 13\* at 2, 4 and 6 months or 2, 3 and 4 months, either 2 doses of *Infanrix hexa* co-administered with *Prevenar* 13 at 3 and 5 months or 2 and 4 months, depending on the immunisation schedule of the country.
  - \*In some countries/regions with an *Infanrix hexa* 3 doses routine national immunisation schedule, *Prevenar* 13 could be administered as 2-doses or 3-doses primary vaccination schedule (according to the routine national immunisation schedule).
- Treatment allocation: non-randomised. All subjects will receive *Infanrix hexa* coadministered with *Prevenar* 13.
- Blinding: Open-label. Note: The study personnel operating GSK Biologicals' randomisation system on internet (SBIR) and the site staff will remain blinded towards the treatment allocation to subjects in study 116945 [DTPA (BOOSTRIX)-047].
- The blinding of study epoch is presented in Table 3.

Table 3 Blinding of study epoch

| Study Epoch | Blinding |
|-------------|----------|
| Epoch 001 | open |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

- Sampling schedule: Blood samples will be drawn from all subjects at the following timepoints:
  - Pre-Pri: Before the first *Infanrix hexa* vaccine administration, a volume of approximately 2 mL of whole blood (to provide approximately 0.7 mL of serum) will be collected from all study participants.
  - Post-Pri: One month after the last dose of *Infanrix hexa* primary vaccination, approximately 5 mL of whole blood (to provide approximately 1.7 mL of serum) will be collected from all study participants.
- Type of study: extension of other protocol(s) 116945 [DTPA (BOOSTRIX)-047].
- Data collection: Electronic Case Report Form (eCRF).
- Safety monitoring: An independent data monitoring committee (IDMC) (including paediatrician and statistician) will be put in place to oversee the safety of infants born to mothers who were vaccinated with Boostrix during pregnancy in the clinical study 116945 [DTPA (BOOSTRIX)-047] i.e. each SAE/incidence of grade 3 local and general solicited AEs, unsolicited AEs will be reviewed by this committee as per IDMC approved charter.

## 3. OBJECTIVES

## 3.1. Primary objective

• To assess the immunological response to *Infanrix hexa* in terms of seroprotection status for diphtheria, tetanus, hepatitis B, poliovirus and Hib antigens, and in terms of vaccine response to the pertussis antigens, one month after the last dose of the primary vaccination in infants born to mothers vaccinated with Boostrix during pregnancy or immediately post-delivery.

Refer to Section 4.1 for the definition of the primary endpoint.

## 3.2. Secondary objectives

- To assess persistence of antibodies against diphtheria, tetanus and pertussis antigens, before the first dose of *Infanrix hexa* in infants born to mothers vaccinated with Boostrix during pregnancy or immediately post-delivery.
- To assess the immunological response to *Infanrix hexa* and *Prevenar 13* in terms of antibody concentrations or titres against all antigens, one month\* after the last dose of the primary vaccination in infants born to mothers vaccinated with Boostrix during pregnancy or immediately post-delivery.
- To assess the immunological response to *Infanrix hexa* in terms of seropositivity rates against pertussis antigens, one month after the last dose of the primary vaccination in infants born to mothers vaccinated with Boostrix during pregnancy or immediately post-delivery.
- To assess the safety and reactogenicity of *Infanrix hexa* and *Prevenar 13* in terms of solicited and unsolicited symptoms and serious adverse events (SAEs).
  - \*In some countries/regions with an *Infanrix hexa* 3-dose vaccination schedule, *Prevenar* 13 could be administered as 2-doses or 3-doses primary vaccination schedule (according to the routine national immunisation schedule). In such an instance, the evaluation will be performed one month after the last *Infanrix hexa* dose regardless of *Prevenar* 13 vaccination. In the countries/regions with an *Infanrix hexa* 2-dose schedule, *Prevenar* 13 is co-administered at the same time as *Infanrix hexa*.

Refer to Section 4.2 for the definition of the secondary endpoints.

#### 4. ENDPOINTS

## 4.1. Primary endpoints

- Immunogenicity with respect to components of *Infanrix hexa*.
  - Anti-diphtheria, anti-tetanus, anti-HBs, anti-poliovirus type 1, anti-poliovirus type 2, anti-poliovirus type 3 and anti-polyribosyl-ribitol phosphate (anti-PRP) seroprotection status, one month after the last dose of primary vaccination.

A seroprotected subject is a subject whose antibody concentration/titre is greater than or equal to the level defining clinical protection. The following seroprotection thresholds are applicable:

- Anti-diphtheria antibody concentrations  $\ge$  0.1 IU/mL.
- Anti-tetanus antibody concentrations  $\geq 0.1 \text{ IU/mL}$ .
- Anti-HBs antibody concentrations  $\ge 10 \text{ mIU/mL}$ .
- Anti-poliovirus types 1, 2 and 3 antibody titres  $\geq 8$ .
- Anti-PRP antibody concentrations  $\geq 0.15 \,\mu g/mL$ .
- Vaccine response to PT, FHA and PRN antigens, one month after the last dose of primary vaccination.

Vaccine response to the PT, FHA and PRN antigens, is defined as:

- appearance of antibodies in subjects who were initially seronegative (i.e., with concentrations <cut-off value).</li>
- at least maintenance of pre-vaccination antibody concentrations in subjects who were initially seropositive (i.e., with concentrations ≥cut-off value).

## 4.2. Secondary endpoints

- Persistence of antibodies before the first dose of Infanrix hexa.
  - Anti-diphtheria and anti-tetanus seroprotection status, anti-PT, anti-FHA, anti-PRN seropositivity status and antibody concentrations.
- Immunogenicity with respect to components of *Infanrix hexa* and Prevenar 13.
  - Anti-diphtheria, anti-tetanus, anti-poliovirus type 1, anti-poliovirus type 2, anti-poliovirus type 3, anti-HBs, anti-PRP, anti-PT, anti-FHA, anti-PRN and anti-pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) antibody concentrations or titres, one month after the last dose of primary vaccination.
- Immunogenicity with respect to components of *Infanrix hexa*.
  - Anti-PT, anti-FHA, anti-PRN antibody seropositivity status, one month after the last dose of primary vaccination.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

- Solicited local and general symptoms.
  - Occurrence of solicited local/general symptoms during the 4-day (Day 0-Day 3) follow-up period after each vaccination.
- Unsolicited adverse events.
  - Occurrence of unsolicited symptoms during the 31-day (Day 0-Day 30) follow-up period after each vaccination.
- Serious adverse events.
  - Occurrence of SAEs from first vaccination dose to study end.

### 5. ANALYSIS SETS

#### 5.1. Definition

## 5.1.1. All enrolled subjects

 All subjects for whom study invasive procedure has been achieved and informed consent has been obtained.

## 5.1.2. Total vaccinated cohort (TVC)

The TVC will include all vaccinated subjects for whom data are available.

- A safety analysis based on the TVC will include all subjects with at least one vaccine administration documented.
- An immunogenicity analysis based on the TVC will include vaccinated subjects for whom data concerning immunogenicity endpoint measures are available.

## 5.1.3. ATP cohort for analysis of safety

The ATP cohort for analysis of safety will include all subjects from the TVC who complied with the vaccine administration:

- who have received at least one dose of study vaccines according to their random assignment.
- for whom administration route and site of study vaccines is known and according to the protocol.
- who have not received a vaccine not specified or forbidden in the protocol.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## 5.1.4. ATP cohort for analysis of immunogenicity

The ATP cohort for immunogenicity will include all evaluable subjects from the ATP cohort for safety:

- who meet all eligibility criteria;
- who comply with the procedures and intervals defined in the protocol.
- who do not meet any of the criteria for elimination from an ATP analysis (refer to Section 6.7.2 of the protocol) during the study;
- who do not receive a product leading to exclusion from an ATP analysis as listed in Section 6.7.2 of the protocol;
- who do not present with a medical condition leading to exclusion from an ATP analysis as listed in Section 6.8 of the protocol;
- who are born full term (full term is defined  $\geq$  37 weeks of gestation);
- for whom data concerning immunogenicity endpoint measures are available. This will include subjects for whom assay results are available for antibodies against at least one study vaccines antigen component.

The interval between the last vaccination visit and post-primary blood sampling, considered for inclusion of a subject will be 21–48 days.

## 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

## 5.2.1. Elimination from Total vaccinated cohort (TVC)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraud data) will be used for identifying subjects eliminated from TVC.

## 5.2.2. Elimination from ATP cohort for safety

#### 5.2.2.1. Excluded subjects

All eliminations from the primary study 116945 [DTPA(BOOSTRIX)-047] will be applicable for this follow up study except for the visit specific elimination codes (2090, 2100 and 2120) in other words the code 1050, 1060, 1070 assigned to the mother in study 116945 [DTPA(BOOSTRIX)-047] will be inherited to the infant.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

A subject will be excluded from the ATP cohort for safety and immunogenicity under the following conditions

| Code | Decode => Condition under which the code is used |
|---|---|
| 900 | Questionable subject => Invalid informed consent or fraudulent data. In case informed consent is obtained retrospectively the subject is not eliminated. |
| 1030 | Study vaccine dose not administered at all but subject number allocated => subjects enrolled but not vaccinated |
| 1040 | Administration of vaccine(s) forbidden in the protocol Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device). A vaccine not foreseen by the study protocol administered during the period starting from 30 days before each dose of vaccine and ending 30 days after*, with the exception of inactivated influenza vaccine and other vaccines given as a part of the national/regional immunisation schedule, that are allowed at any time during the study period. *In case an emergency mass vaccination for an unforeseen public health threat (e.g.: a pandemic) is organised by the public health authorities, outside the routine immunisation program, the time period described above can be reduced if necessary for that vaccine provided it is licensed and used according to its SPC or package insert (PI) and according to the local governmental recommendations and provided a written approval of the Sponsor is obtained. |
| 1050 | Randomisation failure (subject who received a vaccine not compatible with randomization) This code is inherited from the mother. |
| 1060 | Randomisation code broken at the investigator site OR at GSK Safety department. This code is inherited from the mother. |
| 1070 | Incomplete vaccination course before treatment withdrawal: =>for instance only part of the multiple planned administrations at one visit has been administered. For instance, Prevenar not administered while <i>Infanrix hexa</i> is. when no study vaccination at a visit, no other study vaccination can occur up to conclusion/drop-out (Ex. No vaccination at visit 2, but vaccinations at visits 1 and 3 would lead to assignment of code 1070). Note that the code would not be proposed for a subject who had vaccination as planned but missed the last vaccination(s) due to drop-out. In the example given previously, the code would not be proposed if the subject had missed also the vaccination at visit 3). This code is also inheritated from the mother Site or route of study vaccine administration wrong or unknown. Vaccine temperature deviation (vaccine administration not as per protocol) => <i>Infanrix hexa</i> vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation |
| 1090 | Expired vaccine administered (vaccine administration not as per protocol)=> Subjects who received an expired Infanrix hexa |

## 5.2.3. Elimination from ATP cohort for immunogenicity

## 5.2.3.1. Excluded subjects

All eliminations from the primary study 116945 [DTPA(BOOSTRIX)-047] will be applicable for this follow up study except for the visit specific elimination codes (2090, 2100 and 2120).

A subject will be excluded from the ATP cohort for immunogenicity when he/she is excluded from the ATP cohort for safety (see Section 5.1.3)

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

The following additional codes will be used:

| Code | Decode => Condition under which the code is used |
|---|---|
| 2010 | Protocol violation (inclusion/exclusion criteria) including age and excluding codes |
| | mentioned below. |
| | A male or female between, 6 and 14 weeks of age (including 6 weeks and up to and |
| | including 14 weeks and 6 days of age) at the time of the first vaccination. |
| | Healthy subjects as established by medical history and clinical examination before entering |
| | into the study. |
| | This code is also inheritated from the mother |
| 2040 | Administration of any medication forbidden by the protocol=> |
| | Immunosuppressants or other immune-modifying drugs administered chronically (i.e. more |
| | than 14 days) since birth. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, |
| | or equivalent. Inhaled and topical steroids are allowed. |
| | Long-acting immune-modifying drugs administered at any time during the study period |
| | (e.g. infliximab). |
| | This code is also inheritated from the mother |
| 2050 | Underlying medical condition forbidden by the protocol => |
| | Subjects may be eliminated from the ATP cohort for immunogenicity if, during the study, |
| | they incur a condition that has the capability of altering their immune response (e.g. any |
| | confirmed or suspected immunosuppressive or immunodeficient condition) or are |
| | confirmed to have an alteration of their initial immune status. |
| 2080 | Vaccination done but: noncompliance with vaccination schedules (dates of vaccination not |
| | corresponding to protocol intervals or unknown vaccination dates) |
| | Intervals between study visits for subjects vaccinated with <i>Infanrix hexa</i> at 2, 4 and 6 |
| | months of age is 42-104 days from birth to visit 1, 52-78 days from visit 1 to visit 2, 52-78 |
| | days from visit 2 to visit 3. |
| | Intervals between study visits for subjects vaccinated with <i>Infanrix hexa</i> at 2, 3 and 4 |
| | months of age is 42-104 days from birth to visit 1, 21-48 days from visit 1 to visit 2, 21-48 |
| | days from visit 2 to visit 3. |
| | Intervals between study visits for subjects vaccinated with <i>Infanrix hexa</i> at 2 and 4 months |
| | of age is 42 to 104 days from birth to visit 1, 52-78 days from visit 1 to visit 2. |
| | Intervals between study visits for subjects vaccinated with Infanrix hexa at 3 and 5 months |
| | of age is 42 to 104 days from birth to visit 1, 52-78 days from visit 1 to visit 2. |
| 2090 | Blood sample taken but: noncompliance with blood sampling schedules (dates of blood |
| 2030 | sampling not corresponding to adapted protocol intervals or unknown blood |
| | sample/vaccination dates) => 21-48 days from last vaccination visit to visit 4 |
| | Sample/vaccination dates) => 21-40 days from last vaccination visit to visit 4 |
| 0400 | October 19 and 1 |
| 2100 | Serological results not available for antigens POST vaccination (including lost samples, |
| | blood sample not done, unable to test, absence of parallelism) => no immunogenicity |
| 2122 | results available at visit 4. |
| 2120 | Obvious incoherence, abnormal serology evolution or error in data (incoherence between |
| | CRF and results, wrong sample labelling) |

## 6. STATISTICAL ANALYSES

Note that standard data derivation rule and stat methods are described in annex 1 (see Section 11) and will not be repeated below.

## 6.1. Demography

## 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age in weeks, race, height [cm], weight [kg], head circumference [cm], body mass index in [kg/m²]), cohort description and withdrawal status will be summarised by group using descriptive statistics:

- Frequency tables will be generated for categorical variables such as race;
- Mean, median and standard deviation will be provided for continuous data such as age.

The distribution of subjects enrolled among the study sites will be tabulated as a whole and per group.

#### 6.1.2. Additional considerations

Gender, country, schedule of vaccination will also be summarised by group using above mentioned descriptive statistics.

All demography summaries will be generated for the TVC. The summary of age, height, weight, head circumference, gender will also be provided for the ATP cohort for immunogenicity.

Number and reason for elimination from ATP cohorts will be tabulated by group.

Quartile 1 and quartile 3 will be provided for continuous data such as age in weeks, race, height [kg], head circumference [cm], body mass index in [kg/m²].

## 6.2. Exposure.

### 6.2.1. Analysis of exposure planned in the protocol

NA

#### 6.2.2. Additional considerations

The number of doses administered will be summarized by vaccine.

## 6.3. Immunogenicity

## 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be based on the ATP cohort for analysis of immunogenicity. If in any vaccine group, the percentage of enrolled subjects excluded from this ATP cohort is more than 5%, a second analysis based on the TVC will be performed to complement the ATP analysis. All analyses will be descriptive. For each group, at each timepoint that a blood sample result is available:

- Seropositivity rates against PT, FHA and PRN antigens and pneumococcal antigens (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) with exact 95% CI [Clopper, 1934] will be calculated.
- Seroprotection rates against diphtheria toxoid, tetanus toxoid, HBs, PRP antigen and poliovirus types 1, 2, 3 antigens (with exact 95% CI [Clopper, 1934]) will be calculated.
- Percentage of subjects with anti-pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F) antibody concentrations, depending on the GSK laboratory or WHO reference laboratory assay cut-offs, will be calculated along with its exact 95% CI [Clopper, 1934].
- Percentage of subjects with anti-D and anti-T antibody concentrations ≥ 1.0 IU/mL will be calculated along with its exact 95% CI [Clopper, 1934].
- Percentage of subjects with anti-PRP antibody concentrations ≥ 1.0 µg/mL and anti-HBs antibody concentrations ≥ 100 mIU/mL will be calculated along with its exact 95% CI [Clopper, 1934].
- GMC/GMT with 95% CI will be tabulated for antibodies against each antigen.

For serology results one month after last vaccination dose:

- The vaccine response rates to PT, FHA and PRN (with exact 95% CI) will be calculated.
- The distribution of antibody concentrations/titres for each antigen will be displayed using reverse cumulative distribution curves (RCCs).
- The distribution of antibody concentrations or titres of each antigen will be tabulated. Additional summaries will be provided based on country.

#### Handling of missing data:

For a given subject and a given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

#### 6.3.2. Additional considerations

Considering that RCC are available and the percentage of subjects with titres/concentration above key thresholds are available, the distribution of antibody concentrations or titres of each antigen will not be tabulated.

In addition to the percentage of seroprotected or seropositive subjects, the percentage of subjects above the following cut-off will be summarized

- Anti-PRP antibody concentrations  $\geq 1.0 \,\mu g/mL$ .
- Anti-diphtheria antibody concentrations ≥ 1.0 IU/mL.
- Anti-tetanus antibody concentrations  $\geq 1.0 \text{ IU/mL}$ .
- Anti-HBs antibody concentrations ≥ 100 mIU/mL.
- Anti-pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, 23F)
   ≥ 0.35 μg/mL.

In light of the number of subjects enrolled in each country, the analysis by country will be replaced with analysis by schedule (2 doses ie 2,4 months combined with 3,5 months versus 3 doses i.e. 2,3,4 months combined with 2,4,6 months).

In addition subgroups analysis according to gestational age (27-32 weeks and 33-36 weeks) and age of the mother (18-24 year, 25-34 year and 35-45 year) will be performed.

The sub-group analyses will be limited to descriptive tables of GMT/GMC and the percentage of subjects with titres/concentration above key thresholds for ATP cohort of immunogenicity.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

| SCHEDULE_TXT(Element Text) country(CTY_NAM) | | | | | | | |
|---|---|---|---|---|---|---|---|
| Frequency<br>Percent<br>Row Pct<br>Col Pct | Australi<br>a | Canada | Czechia | Finland | Italy | Spain | Total |
| Age group(2, 3,<br>4 Months) | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 71<br>11.81<br>100.00<br>100.00 | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 71<br>11.81 |
| Age group(2, 4 M<br>onths) | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 7<br>1.16<br>100.00<br>2.48 | 7<br>1.16 |
| Age group(2, 4,<br>6 Months) | 38<br>6.32<br>8.32<br>100.00 | 144<br>23.96<br>31.51<br>100.00 | 0.00<br>0.00<br>0.00 | 0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 275<br>45.76<br>60.18<br>97.52 | 457<br>76.04 |
| Age group(3, 5 M<br>onths) | 0.00<br>0.00<br>0.00 | 0<br>0.00<br>0.00<br>0.00 | 0.00<br>0.00<br>0.00 | 52<br>8.65<br>78.79<br>100.00 | 14<br>2.33<br>21.21<br>100.00 | 0.00<br>0.00<br>0.00 | 66<br>10.98 |
| Total | 38<br>6.32 | 144<br>23.96 | 71<br>11.81 | 52<br>8.65 | 14<br>2.33 | 282<br>46.92 | 601<br>100.00 |

Deviations from specifications for age and intervals between study visits for subjects vaccinated with *Infanrix hexa* by dose schedule (2 dose schedule and 3 dose schedule separately) will be tabulated.

## 6.4. Analysis of safety

## 6.4.1. Analysis of safety and reactogenicity planned in the protocol

The primary analysis will be based on the TVC. If more than 5% of enrolled subjects are excluded from the ATP cohort for analysis of safety, then a second analysis based on this ATP cohort will be performed to complement the TVC analysis. All analyses will be descriptive.

• The percentage of doses and of subjects with at least one local symptom (solicited or unsolicited), with at least one general symptom (solicited or unsolicited) and with any symptom (solicited or unsolicited) during the 4-day (Day 0-Day 3) solicited follow-up period will be tabulated with exact 95% CI [Clopper, 1934] after each vaccine dose and overall. The same calculations will be done for symptoms (solicited or unsolicited) rated as grade 3 in intensity, for symptoms (solicited or unsolicited) leading to medical advice and for symptoms (solicited or unsolicited) assessed as causally related to vaccination.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

- The percentage of doses and of subjects reporting each individual solicited local and general symptom during the 4-day (Day 0-Day 3) solicited follow-up period will be tabulated after each vaccine dose and overall, with exact 95% CI [Clopper, 1934]. The same calculations will be done for each individual solicited symptom rated as grade 3 in intensity and for each individual solicited symptom assessed as causally related to vaccination.
- All computations mentioned above will be done for grade ≥2 (solicited symptoms only) and grade 3 symptoms, for symptoms considered related to vaccination (general symptoms only) and for symptoms that resulted in a medically-attended visit
- Occurrence of fever and related fever will be reported per 0.5°C cumulative temperature increments as well as the occurrence of grade 3 fever (> 39.0°C axillary temperature) with causal relationship to vaccination.
- The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to MedDRA. Every verbatim term will be matched with the appropriate Preferred Term. The percentage of subjects with unsolicited AEs occurring within 31-day (Day 0- Day 30) follow-up period after any dose with its exact 95% CI [Clopper, 1934] will be tabulated by group, and by preferred term. Similar tabulation will be done for unsolicited AEs rated as grade 3, for unsolicited AEs with causal relationship to vaccination and AEs/SAEs leading to withdrawal from the study.
- The percentage of subjects who receive concomitant medication and antipyretic medication during the 4-day (Day 0- Day 3) follow-up period and the 31-day follow-up (Day 0 Day 30) will be tabulated (with exact 95% CI [Clopper, 1934]) after each vaccine dose and overall.
- SAEs reported from first vaccination dose up to study end will be described in detail.
- Withdrawal due to AEs and SAEs following vaccinations will be described in detail.

#### Handling of missing data:

- For a given subject and the analysis of solicited AEs 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited AEs based on the TVC will include only vaccinated subjects and doses with documented safety data (i.e. symptom screen completed).
- For analysis of unsolicited AEs, such as SAEs or AEs by primary Medical Dictionary for Regulatory Activities (MedDRA) term, and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.
- For summaries reporting both solicited and unsolicited AEs, all vaccinated subjects will be considered. Subjects, who do not report the event or the concomitant medication, will be considered as subjects without the event or the concomitant medication, respectively.

#### 6.4.2. Additional considerations

#### 6.4.2.1. Combined Solicited and Unsolicited Adverse Events

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes.

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| PA | 10022086 | Injection site pain |
| RE | 10022098 | Redness at injection site |
| SW | 10053425 | Swelling at injection site |
| TE | 10016558 | Temperature/Fever |
| FU | 10022998 | Irritability/Fussiness |
| DR | 10013649 | Drowsiness |
| LO | 10003028 | Loss of appetite |

## 7. ANALYSIS INTERPRETATION

All analyses will be conducted in a descriptive manner.

#### 8. CONDUCT OF ANALYSES

Any deviation(s) or change(s) from the original statistical plan outlined in this protocol will be described and justified in the final study report.

## 8.1. Sequence of analyses

The final analyses of all data will be conducted when all data are available. This analysis will include the final analysis of immunogenicity and the final analysis of solicited and unsolicited symptoms and SAEs. A clinical study report containing all data will be written and made available to the investigators.

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=public<br>posting, SR=study<br>report, internal,<br>public posting) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference<br>for TFL |
|---|---|---|---|---|---|
| Final | E1_01 | SR | Yes | Yes | TFL TOC |

## 8.2. Statistical considerations for interim analyses

NA

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### 9. CHANGES FROM PLANNED ANALYSES

- During the course of the study, the assays used to measure the anti-D, anti-T, anti-PT, anti-FHA and anti-PRN IgG concentrations were re-developed and re-validated and both assay units and assay cut-offs were adapted. The new ELISA's for PT, FHA and PRN were calibrated against the WHO International Standard (NIBSC 06/140). This allowed the expression of concentrations measured with the new ELISA's in international units per milliliter (IU/mL) instead of the formerly used ELISA units per milliliter (ELU/mL). The newly validated DTPa ELISA's used in the study have a lower assay cut-off as compared to the one described in the protocol. The current assay cut-off is 0.057 IU/mL for anti-D, 0.043 IU/mL for anti-T, 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti- PRN. An agreement between the old and new ELISAs was shown with regards to the two thresholds of clinical relevance for the DI/TE response (0.1 IU/mL and 1.0 IU/mL) and therefore the clinical endpoints and anti-D and anti-T are unchanged. In the absence of a correlate of protection for the B. pertussis antigens, the pertussis endpoints were redefined based on the assay cut-off (see section 5.7.5 of protocol).
- In addition, following CBER feedback on the anti-D re-validated assay, a calibration factor of 0.543 was applied in the analysis of anti-D in order to align the ELISA assay to the WHO 10/262 reference samples which are measured as 2 IU/mL by Di neutralization. Assay since 54 WHO 10/262 reference samples measured by GSK re-validated ELISA led to GMC was about two fold (1.841) higher than the expected value (2 IU/mL).

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

• Note: Due to re-validation of all assays, the cut-offs presented in Table 11 of the protocol of few antigens have changed. Below table has an updated threshold.

| Antigen | Threshold for positivity |
|-------------------------------------|--------------------------|
| • Anti-PT | • 2.693 IU/mL |
| • Anti-FHA | • 2.046 IU/mL |
| • Anti-PRN | • 2.187 IU/mL |
| • Anti-D | • 0.057 IU/mL |
| • Anti-T | • 0.043 IU/mL |
| • Anti-polio | 8 dilution |
| Anti-PRP | • 0.066 μg/mL |
| • Anti-HBs | • 6.2 mIU/mL |
| • Anti-pneumococcal serotypes (1) | • 0.080 μg/mL |
| • Anti-pneumococcal serotypes (3) | • 0.075 μg/mL |
| • Anti-pneumococcal serotypes (4) | • 0.061 μg/mL |
| • Anti-pneumococcal serotypes (5) | • 0.198 μg/mL |
| • Anti-pneumococcal serotypes (6A) | • 0.111 μg/mL |
| Anti-pneumococcal serotypes (6B) | • 0.102 μg/mL |
| • Anti-pneumococcal serotypes (7F) | • 0.063 μg/mL |
| • Anti-pneumococcal serotypes (9V) | • 0.066 μg/mL |
| • Anti-pneumococcal serotypes (14) | • 0.160 μg/mL |
| • Anti-pneumococcal serotypes (18C) | • 0.111 μg/mL |
| • Anti-pneumococcal serotypes (19A) | • 0.199 μg/mL |
| • Anti-pneumococcal serotypes (19F) | • 0.163 μg/mL |
| • Anti-pneumococcal serotypes (23F) | • 0.073 μg/mL |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The TFL TOC (Tables Figures and Listings Table Of Contents) provides the list of tables/listings and figures needed for the study report (synopsis, in-text, post-text) and for public disclosure (CTRS).

The following group names will be used in the TFLs:

| Group<br>order in<br>tables | Group label in tables | Group definition for footnote | Pooled Groups label in tables | Pooled definition for footnote |
|---|---|---|---|---|
| 1 | dTpa Group | Infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047] where mothers received dTpa during pregnancy. All subjects in this group will receive <i>Infanrix hexa</i> coadministered with <i>Prevenar 13</i> according to the routine national immunisation schedule. | NA | NA |
| 2 | Control Group | Infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047] where mothers received placebo during pregnancy. All subjects in this group will receive <i>Infanrix hexa</i> coadministered with <i>Prevenar 13</i> according to the routine national immunisation schedule. | NA | NA |

Tables will be generated on ATP cohort for immunogenicity with the following subgroup names inherited from the study 116945 [DTPA (BOOSTRIX)-047]

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 18-24Y | 18-24 years old subjects |
| 2 | 25-34Y | 25-34 years old subjects |
| 3 | 35-45Y | 35-45 years old subjects |
| 4 | 27-32W | 27-32 weeks of gestation of foetus at dose 1 |
| 5 | 33-36W | 33-36 weeks of gestation of foetus at dose 1 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

#### 11.1. Statistical Method References

- The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. Biometrika. 1934; 26:404-413].
- The 95% CI for geometric mean titers/concentrations (GMTs/GMCs) will be obtained within each group separately. The 95% CI for the mean of log-transformed titer/concentration will be first obtained assuming that log-transformed values were normally distributed with unknown variance. The 95% CI for the GMTs/GMCs will be then obtained by exponential-transformation of the 95% CI for the mean of log-transformed titer/concentration.

#### 11.2. Standard data derivation

#### 11.2.1. Date derivation

- SAS date derived from a character date: In case day is missing, 15 is used. In case day & month are missing, 30 June is used.
- Onset day for an event for the infant (AE, medication, vaccination, ...): The onset day is the number of days from date of last study dose & the onset/start date of the event. This is 0 for an event starting on the same day of last study dose. There could also be events reported in the infant before delivery (anomalies diagnosed during pregnancy at ultrasound investigation), for these cases onset day will be negative '-' days. See SAS date derived in case the start date of the event is incomplete.
- Duration: Duration of an event is expressed in days. It is the number of days between the start & the stop dates + 1. Therefore duration is 1 day for an event starting & ending on the same day.

#### 11.2.2. Dose number

The study dose number is defined in reference to the number of study visits at which vaccination occurred. More specifically dose 1 refers to all vaccines administered at the first vaccination visit while dose 2 corresponds to all vaccinations administered at the second vaccination visit even if this is the first time a product is administered to the subject.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

Relative dose: the relative dose for an event (AE, medication, vaccination) is the most recent study dose given before an event. In case the event takes place on the day a study dose is given, the related dose will be that of the study dose, even if the event actually took place before vaccination. For instance, if an adverse event begins on the day of the study vaccination but prior to administration of the vaccine, it will be assigned to this dose. In case a study dose is not administered and an event occurs after the subsequent study dose (e.g. 3rd study dose), the relative dose of the event will be study dose associated to the subsequent study dose (e.g. dose 3).

The number of doses for a product is the number of time the product was administered to a subject.

The incidence per dose is the number of vaccination visits at which an event (vaccination visit is a visit at which study vaccine was administered) was reported among all vaccination visits.

## 11.2.3. Demography

Age: Age at the reference activity, computed as the number of units between the date of birth and the reference activity.

Conversion of weight to kg

The following conversion rule is used:

Weight in Kilogram= weight in Pounds / 2.2

Weight in Kilogram = weight in oncs / 35.2

The result is rounded to 2 decimals.

Conversion of height to cm

The following conversion rule is used:

Height in Centimetres = Height in Feet \* 30.48

Height in Centimetres = Height in Inch \* 2.54

The result is rounded to the unit (i.e no decimal)

Conversion of temperature to °C

The following conversion rule is used:

Temperature in °Celsius = ((Temperature in °Fahrenheit -32) \*5)/9

The result is rounded to 1 decimal.

## 11.2.4. Immunogenicity

For a given subject and given immunogenicity measurement, missing or non-evaluable measurements will not be replaced. Therefore, an analysis will exclude subjects with missing or non-evaluable measurements.

The Geometric Mean Concentrations/Titres (GMC/Ts) calculations are performed by taking the anti-log of the mean of the log titre transformations. Antibody titres below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

A seronegative subject is a subject whose antibody titre is below the cut-off value of the assay. A seropositive subject is a subject whose antibody titre is greater than or equal to the cut-off value of the assay.

The assay cut-off is the value under which there is no quantifiable result available. For an assay with a specific 'cut\_off', numerical immunogenicity result is derived from a character field (rawres):

```
If rawres is 'NEG' or '-' or '(-)', numeric result= cutt_off/2,

if rawres is 'POS' or '+' or '(+)', numeric result = cut_off,

if rawres is '< value' and value<=cut_off, numeric result = cut_off/2,

if rawres is '< value' and value>cut_off, numeric result = value,

if rawres is '> value' and value<cut_off, numeric result = cut_off/2,

if rawres is '> value' and value>=cut_off, numeric result = value,

if rawres is '<= value' or '>= value' and value<cut_off, numeric result = cut_off/2,

if rawres is '<= value' or '>= value' and value>=cut_off, numeric result = value,

if rawres is a value < cut_off, numeric result = cut_off/2,

if rawres is a value >= cut_off, numeric result = rawres,

if rawres is a value >= cut_off, numeric result = rawres,
```

else numeric result is left blank.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## 11.2.5. Safety

For analysis of solicited, unsolicited adverse events such as serious adverse events or adverse events by primary MedDRA term, and for the analysis of concomitant medications, all vaccinated subjects will be considered. Subjects who did not report the event or the concomitant medication will be considered as subjects without the event or the concomitant medication respectively.

For a given subject and the analysis of solicited adverse events within 4 days post-vaccination, missing or non-evaluable measurements will not be replaced. Therefore, the analysis of the solicited adverse events based on the Total Vaccinated Cohort will include only vaccinated subjects for doses with documented safety data (i.e., symptom screen completed). More specifically the following rules will be used:

- Subjects who documented the absence of a solicited adverse events after one dose will be considered not having that adverse events after that dose.
- Subjects who documented the presence of a solicited symptom and fully or partially recorded daily measurement over the solicited period will be included in the summaries at that dose and classified according to their maximum observed daily recording over the solicited period.
- Subjects who documented the presence of a solicited symptom after one dose without having recorded any daily measurement will be assigned to the lowest intensity category at that dose (i.e., 37.5°C for fever or grade 1 for other symptoms).
- Doses without symptom sheets documented will be excluded.
- The intensity of the following solicited adverse events will be assessed as described in the below table

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

Table 4 Intensity scales for solicited symptoms in infants less than 6 years of age

| Adverse Event | Intensity grade | Parameter |
|---|---|---|
| Pain at injection site | 0 | None |
| - | 1 | Mild: Minor reaction to touch |
| | 2 | Moderate: Cries/protests on touch |
| | 3 | Severe: Cries when limb is moved/spontaneously painful |
| Redness at injection site | | Record greatest surface diameter in mm |
| Swelling at injection site | | Record greatest surface diameter in mm |
| Fever* | | Record temperature in °C/°F |
| Irritability/Fussiness | 0 | Behaviour as usual |
| , | 1 | Mild: Crying more than usual/no effect on normal activity |
| | 2 | Moderate: Crying more than usual/interferes with normal |
| | | activity |
| | 3 | Severe: Crying that cannot be comforted/prevents normal |
| | | activity |
| Drowsiness | 0 | Behaviour as usual |
| | 1 | Mild: Drowsiness easily tolerated |
| | 2 | Moderate: Drowsiness that interferes with normal activity |
| | 3 | Severe: Drowsiness that prevents normal activity |
| Loss of appetite | 0 | Appetite as usual |
| | 1 | Mild: Eating less than usual/no effect on normal activity |
| | 2 | Moderate: Eating less than usual/interferes with normal activity |
| | 3 | Severe: Not eating at all |

<sup>\*</sup>Fever is defined as temperature  $\geq$  37.5°C / 99.5°F for oral, axillary or tympanic route, or  $\geq$  38.0°C / 100.4°F for rectal route. The preferred route for recording temperature in this study will be rectal/axillary.

The maximum intensity of local injection site redness/swelling will be scored at GSK Biologicals as follows:

| 0 | Absent |
|---|--------------------|
| 1 | ≤ 5 mm |
| 2 | > 5 mm and ≤ 20 mm |
| 3 | > 20 mm |

The maximum intensity of fever (oral, axillary or tympanic route) will be scored at GSK Biologicals as follows:

| Grade | Temperature |
|-------|--------------------|
| 0 | <37.5°C |
| 1 | ≥37.5°C to ≤38.0°C |
| 2 | >38.0°C to ≤39.0°C |
| 3 | > 39.0°C |

The investigator will assess the maximum intensity that occurred over the duration of the event for all unsolicited AEs (including SAEs) recorded during the study. The assessment will be based on the investigator's clinical judgement.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

The intensity should be assigned to one of the following categories:

| 1 (mild) | <ul> <li>An AE which is easily tolerated by the subject, causing minimal discomfort and not</li> </ul> |
|---|---|
| | interfering with everyday activities. |
| 2 (moderate) | = An AE which is sufficiently discomforting to interfere with normal everyday activities. |
| 3 (severe) | = An AE which prevents normal, everyday activities (in a young child, such an AE would, |
| | for example, prevent attendance at school/kindergarten/a day-care centre and would |
| | cause the parent(s)/LAR(s) to seek medical advice |

An AE that is assessed as Grade 3 (severe) should not be confused with a SAE. Grade 3 is a category used for rating the intensity of an event; and both AEs and SAEs can be assessed as Grade 3. An event is defined as 'serious' when it meets one of the pre-defined outcomes as described in Section 8.1.2 in the protocol.

The way the percentage of subjects will be derived will depend on the event analysed (see table below for details). As a result, the N value will differ from one table to another.

| Event | N used for deriving % per subject | N used for deriving % per dose |
|---|---|---|
| Concomitant vaccination | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Solicited general AEs | All subjects with at least one solicited general AE documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited general AE documented as either present or absent (i.e., symptom screen completed) |
| Solicited local AEs | All subjects with at least one solicited local AE documented as either present or absent (i.e., symptom screen completed) | All study visits with study vaccine administered and with at least one solicited local AE documented as either present or absent (i.e., AE screen completed) |
| Unsolicited AEs | All subjects with study vaccine administered | All study visits with study vaccine administered |
| Concomitant medication | All subjects with study vaccine administered | All study visits with study vaccine administered |

## 11.2.6. Number of decimals displayed:

The following decimal description from the decision rules will be used for the demography, immunogenicity and safety/reactogenicity.

| Display Table | Parameters | Number of decimal digits |
|---|---|---|
| Demographic characteristics | Mean, median age | 1 |
| Demographic characteristics | SD (age) | 1 |
| Immunogenicity | GMT/GMC | 3 for anti-D, anti-T and anti-PRP 2 for Strepto antigens 1 for anti-PT, anti-FHA and anti-PRN, anti-HBs, anti-Polio 1, anti-Polio 2 and anti-Polio 3 |
| Reactogenicity | Mean, Min, Q1, Median, Q3, Max for duration | 1 |
| All summaries | % of count, including LL & UL of CI | 1 |

## 12. ANNEX 3: STUDY SPECIFIC MOCK TFL

The following drafted study specific mocks will be used.

The data display, title and footnote is for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC.

These templates were copied from recent studies. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

Template 1 Number of subjects enrolled by center (Total vaccinated cohort)

| | dTpa Group | Control group | Total | |
|--------|------------|---------------|-------|---|
| Center | n | N | n | % |
| PPD | | | | |
| All | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

n = number of subjects included in each group or in total for a given center or for all centers

All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## Template 2 Number of subjects enrolled by country (Total vaccinated cohort)

| | dTpa Group | Control group | Total | | |
|-----------|------------|---------------|-------|---|---|
| Country | n | N | n | % | |
| Australia | | | | | |
| Belgium | | | | | |
| Canada | | | | | |
| Czechia | | | | | |
| Finland | | | | | |
| Italy | | | | | - |
| Spain | | | | | - |
| All | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

n = number of subjects included in each group or in total for a given country or for all countries All = sum of all subjects in each group or in total (sum of all groups)

 $% = n/AII \times 100$ 

## Template 3 Number of subjects vaccinated, completed and withdrawn with reason for withdrawal (Total vaccinated cohort)

| | dTpa Group | Control<br>Group | Total |
|---|---|---|---|
| Number of subjects vaccinated | | | |
| Number of subjects completed | | | |
| Number of subjects withdrawn | | | |
| Reasons for withdrawal: | | | |
| Serious Adverse Event | | | |
| Non-serious adverse event | | | |
| Protocol violation | | | |
| Consent withdrawal (not due to an adverse event) | | | |
| Migrated/moved from study area | | | |
| Lost to follow-up (subjects with incomplete vaccination course) | | | |
| Lost to follow-up (subjects with complete vaccination course) | | | |
| Others | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Vaccinated = number of subjects who were vaccinated in the study

Completed = number of subjects who completed last study visit

Withdrawn = number of subjects who did not come for last study visit
201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 4 Number of subjects at each visit and list of withdrawn subjects (Total Vaccinated Cohort)

| Group | VISIT | N | Withdrawn Subject | Reason for withdrawal |
|---|---|---|---|---|
| dTpa Group | VISIT 1 | 508 | | |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 504 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | SERIOUS ADVERSE EXPERIENCE |
| | VISIT 3 | 501 | | |
| | | | no. P | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| | | | no. PPD | MIGRATION FROM STUDY AREA |
| Control<br>Group | VISIT 1 | 257 | | |
| | | | no. PP | PROTOCOL VIOLATION |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 2 | 255 | | |
| | | | no. PPD | CONSENT WITHDRAWAL |
| | VISIT 3 | 254 | | |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PP | LOST TO FOLLOW-UP |
| | | | no.PPD | LOST TO FOLLOW-UP |
| | | | no. PP | CONSENT WITHDRAWAL |
| | | | no. PP | MIGRATION FROM STUDY AREA |
| | | | no. PPD | LOST TO FOLLOW-UP |
| | | | no. PPD | ADVERSE EXPERIENCE |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = number of subjects who are still in the study up to the visit

Withdrawn = subject who did not return after the visit

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 5 Number of subjects enrolled into the study as well as excluded from ATP analyses with reasons for exclusion

| | Total | | | | dTp:<br>Grou | ıp | | Cont<br>Grou | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Title | N | n | S | % | N | n | S | N | n | S |
| Total enrolled cohort | 1200 | | | | 300 | | | 300 | | |
| Invalid informed consent or fraud data (code 900) | | | | | | | | | | |
| Study vaccine dose not administered AT ALL but subject number allocated (code 1030) | | | | | | | | | | |
| TVC | 1200 | | | 100 | 300 | | | 300 | | |
| Administration of vaccine(s) forbidden in the protocol (code 1040) | | 2 | 2 | | | 0 | 0 | | 0 | 0 |
| Randomisation code broken at the investigator site OR at GSK Safety department (1060) | | | | | | | | | | |
| Study vaccine dose not administered according to protocol (code 1070) | | 73 | 73 | | | 23 | 23 | | 16 | 16 |
| Vaccine temperature deviation (code 1080) | | | | | | | | | | |
| Expired vaccine administered (code 1090) | | 10 | 11 | | | 3 | 3 | | 1 | 1 |
| Protocol violation (inclusion/exclusion criteria) (code 2010) | | 1 | 1 | | | 1 | 1 | | 0 | 0 |
| Administration of any medication forbidden by the protocol (code 2040) | | 1 | 1 | | | 0 | 0 | | 1 | 1 |
| Underlying medical condition forbidden by the protocol (code 2050) | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| Concomitant infection related to the vaccine which may influence | | | | | | | | | | |
| immune response (2060) | | | | | | | | | | |
| Concomitant infection not related to the vaccine which may influence immune response (code 2070) | | 0 | 1 | | | 0 | 0 | | 0 | 1 |
| Noncompliance with vaccination schedule (including wrong and unknown dates) (code 2080) | | 14 | 16 | | | 6 | 7 | | 3 | 4 |
| Noncompliance with blood sampling schedule (including wrong and unknown dates) (code 2090) | | 12 | 16 | | | 3 | 5 | | 4 | 5 |
| Essential serological data missing (code 2100) | | 87 | 95 | | | 20 | 22 | | 23 | 26 |
| Obvious incoherence, abnormal serology evolution or error in data (code 2120) | | 1 | 1 | | | 0 | 0 | | 0 | 0 |
| ATP cohort for analysis of immunogenicity | 998 | | | 83.2 | 244 | | | 252 | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Note: Subjects may have more than 1 elimination code assigned

n = number of subjects with the elimination code assigned excluding subjects who have been assigned a lower elimination code number

s = number of subjects with the elimination code assigned

% = percentage of subjects in the per protocol set (ATP) relative to the TVC(ES)

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 6 Deviations from specifications for age and intervals between study visits for subjects vaccinated with Infanrix hexa(<2> dose schedule - 1 dose/visit) (Total Vaccinated Cohort)

| | | Age | VAC:1-VAC:2 | VAC:2-SER:2 |
|---|---|---|---|---|
| Group | | Protocol | Protocol | Protocol |
| | | from 6 to 14 weeks and 6 | from 52 to 78 days | from 21 to 48 days |
| | | days | | , |
| dTpa Group | N | | | |
| | n | | | |
| | % | | | |
| | range | | | |
| Control Group | N | | | |
| · | n | | | |
| | % | | | |
| | range | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = total number of subjects with available results

n(%) = number(percentage) of subjects with results outside of the interval

range = minimum-maximum for age and intervals

VAC:1 = vaccination at visit 1

VAC:2 = vaccination at visit 2

SER:2 = blood sample collected before the first dose and 1 month after the last dose of the primary vaccination course 2 dose schedule = subjects who received 2 dose of *Infanrix hexa* at 2,4 months of age or 3,5 months of age, co-administered with *Prevenar 13* (according to the routine national immunisation schedule of the country).

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 7 Summary of demographic characteristics (Total vaccinated cohort)

| | | dTpa Gro<br>N = | oup | Control G | roup | N = | |
|---|---|---|---|---|---|---|---|
| Characteristics | Parameters or Categories | Value or n | % | Value or<br>n | % | Value or n | % |
| Age (week) at vaccination dose: 1 | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | Q1 | | | | | | |
| | Q3 | | | | | | |
| Gender | Female | | | | | | |
| | Male | | | | | | |
| Geographic Ancestry | African Heritage / African American | | | | | | |
| | American Indian or Alaskan Native | | | | | | |
| | Asian - Central / South Asian | | | | | | |
| | Heritage | | | | | | |
| | Asian - East Asian Heritage | | | | | | |
| | Asian - Japanese Heritage | | | | | | |
| | Asian - South East Asian Heritage | | | | | | |
| | Native Hawaiian or Other Pacific Islander | | | | | | |
| | White - Arabic / North African<br>Heritage | | | | | | |
| | White - Caucasian / European | | | | | | |
| | Heritage<br>Other (Hispanic) | | | | | | |
| Dose schedule | 2 dose schedule | | | | | | |
| DOSE SCHEAMIE | 3 dose schedule | | | | | | |
| Maternal ago group | 18-24Y | | | | | | |
| Maternal age group | 25-34Y | | | | | | |
| | 35-45Y | | | | | | |
| Contational weak of facture of | 27-32W | | | | | | |
| Gestational week of foetus at | 33-36W | | | | | | |
| dose 1 | 33-3011 | | | | | l | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = total number of subjects

n(%) = number(percentage) of subjects in a given category

Value = value of the considered parameter

SD = standard deviation

Q1 = Quartile 1

Q2 = Quartile 3

2 dose schedule = subjects who received 2 dose of Infanrix hexa at 2,4 months of age or 3,5 months of age, co-administered with Prevenar 13 (according to the routine national immunisation schedule of the country).

3 dose schedule = subjects who received 3 dose of Infanrix hexa at 2,3,4 months of age or 2,4,6 months of age, co-administered with Prevenar 13.Prevenar 13 could be administered as 2-doses or 3-doses primary vaccination schedule (according to the routine national immunisation schedule of the country).

18-24Y = 18-24 years old subjects

25-34Y = 25-34 years old subjects

35-45Y = 35-45 years old subjects

27-32W = 27-32 weeks of gestation of foetus at dose 1

33-36W = 33-36 weeks of gestation of foetus at dose 1

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 8 Summary of vital signs characteristics (Total Vaccinated Cohort)

| | | dTpa Group<br>(N = 335) | Control Group<br>(N = 336) | Total<br>(N = 671) |
|---|---|---|---|---|
| Characteristics | Parameters | Value ` | Value | Value |
| Height (cm) | Mean | | | |
| , | SD | | | |
| | Median | | | |
| | Q1 | | | |
| | Q3 | | | |
| | Unknown | | | |
| Weight (kg) | Mean | | | |
| | SD | | | |
| | Median | | | |
| | Q1 | | | |
| | Q3 | | | |
| | Unknown | | | |
| Head circumference (cm) | Mean | | | |
| , , | SD | | | |
| | Median | | | |
| | Q1 | | | |
| | Q3 | | | |
| | Unknown | | | |
| Body mass index in | Mean | | | |
| [kg/m2] | SD | | | |
| | Median | | | |
| | Q1 | | | |
| | Q3 | | | |
| | Unknown | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = total number of subjects

Value = value of the considered parameter

SD = standard deviation

Height (cm) = height expressed in centimeters

Weight (kg) = weight expressed in kilograms

Head circumference(cm) = head circumference expressed in centimeters.

Body mass index in [kg/m2] = body mass index expressed in kilograms per meter square

SD = standard deviation

Q1 = Quartile 1

Q2 = Quartile 3

### Template 9 Study population (TVC)

| Study population (Total vaccinated cohort) | | |
|---|---|---|
| Number of subjects | dTpa group | Control group |
| Planned, N | 225 | 225 |
| Randomised, N (Total Vaccinated Cohort) | 224 | 227 |
| Completed, n (%) | 224 (100) | 227 (100) |
| Demographics | dTpa group | Control group |
| N (Total Vaccinated Cohort) | 224 | 227 |
| Females: Males | 97:127 | 115:112 |
| Mean Age, weeks (SD) | 8.8 (1.1) | 8.8 (1.1) |
| Median Age, weeks (minimum, maximum) | 9 (7, 11) | 9 (7, 11) |
| Most frequent race: Asian - East Asian Heritage, n (%) | 224 (100) | 226 (99.6) |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = total number of subjects enrolled in the study

n/% = number/percentage of subjects in a given category

SD = Standard Deviation

Mean Age = age calculated from Date of birth to first study vaccination

Template 10 Seropositivity rates and GMCs for anti-PT, anti-FHA and anti-PRN antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity)

| | | | | | ≥a | ssay cu | t-off* | | GMC | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 9: | 5% CI |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL |
| Anti-PT | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control Group | Pre-Pri | | | | | | | | |
| | · | Post-Pri | | | | | | | | |
| Anti-FHA | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control Group | Pre-Pri | | | | | | | | |
| | · | Post-Pri | | | | | | | | |
| Anti-PRN | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control Group | Pre-Pri | | | | | | | | |
| | · | Post-Pri | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

\*Assay cut-off is 2.693 IU/mL for anti- PT, 2.046 IU/mL for anti-FHA and 2.187 IU/mL for anti-PRN

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n(%)=number(percentage) of subjects with antibody concentrations above the specified cut-off

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-Pri = blood sample to be collected before the first dose of the primary vaccination course

Post-Pri = blood sample to be collected 1 month after the last dose of the primary vaccination course

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## Template 11 Seropositivity, seroprotection and GMC rates for <anti-tetanus> antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity)

| | | | | ≥ 8 | assa | y cut- | | | ≥ 0.1 | | | ì | ≥ 1.0 | | | | GMC | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | | | 95% CI | | 95% CI | | | 95% | 95% CI | | |
| Antibody | Group | Timing | N | n | % | LL | UL | n | % | LL | UL | n | % | UL | UL | value | LL | UL |
| Anti-<br>tetanus | dTpa<br>Group | Pre-Pri | | | | | | | | | | | | | | | | |
| | ' | Post-Pri | | | | | | | | | | | | | | | | |
| | Control<br>Group | Pre-Pri | | | | | | | | | | | | | | | | |
| | | Post-Pri | | | | | | | | | | | | | | | | |
| Anti-<br>diphtheria | dTpa<br>Group | Pre-Pri | | | | | | | | | | | | | | | | |
| · | | Post-Pri | | | | | | | | | | | | | | | | |
| | Control<br>Group | Pre-Pri | | | | | | | | | | | | | | | | |
| | | Post-Pri | | | | | | | | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

\*Assay cut-off is 0.043 IU/mL for anti-tetanus and 0.057 IU/mL for anti- diphtheria

GMC = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n(%)=number(percentage) of subjects with antibody concentrations above the specified cut-off

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-Pri = blood sample to be collected before the first dose of the primary vaccination course

Post-Pri = blood sample to be collected 1 month after the last dose of the primary vaccination course

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## Template 12 Seroprotection rates for anti-poliovirus type 1,2,3 antibodies before the first dose and 1 month after the last dose of the primary vaccination (ATP cohort for immunogenicity)

| • | | • | | | | ≥8 | | | GMT | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 9: | 5% CI | | 9 | 5% CI |
| Antibody | Group | Timing | N | n | % | UL | UL | value | LL | UL |
| anti-poliovirus type 1 | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control<br>Group | Pre-Pri | | | | | | | | |
| | · · | Post-Pri | | | | | | | | |
| anti-poliovirus type 2 | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control | Pre-Pri | | | | | | | | |
| | Group | Post-Pri | | | | | | | | |
| anti-poliovirus type 3 | dTpa Group | Pre-Pri | | | | | | | | |
| | | Post-Pri | | | | | | | | |
| | Control<br>Group | Pre-Pri | | | | | | | | |
| | ' | Post-Pri | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

GMT = geometric mean antibody concentration calculated on all subjects

N = number of subjects with available results

n(%)=number(percentage) of subjects with antibody concentrations above the specified cut-off

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Pre-Pri = blood sample to be collected before the first dose of the primary vaccination course

Post-Pri = blood sample to be collected 1 month after the last dose of the primary vaccination course

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 13 Vaccine responses for anti-PT, anti-FHA and anti-PRN antibody concentration 1 month after the last dose of the primary vaccination course (ATP cohort for immunogenicity)

| | | | | | Vacci | ne respo | nse |
|---|---|---|---|---|---|---|---|
| | | | | | | | 5% CI |
| Antibody | Group | Pre-Pri*<br>status | N | n | % | LL | UL |
| anti-PT | dTpa Group | S- | | | | | |
| | | S+ (≥cut-off IU/mL)<br>Total | | | | | |
| | Control Group | S- | | | | | |
| | | S+ (≥cut-off IU/mL) | | | | | |
| anti-FHA | dTpa Group | Total<br>S- | | | | | |
| | | S+ (≥cut-off IU/mL) | | | | | |
| | Control Croup | Total<br>S- | | | | | |
| | Control Group | S+ (≥cut-off IU/mL) | | | | | |
| | | Total | | | | | |
| anti-PRN | dTpa Group | S- | | | | | |
| | | S+ (≥cut-off IU/mL)<br>Total | | | | | |
| | Control Group | S- | | | | | |
| | | S+ (≥cut-off IU/mL) | | | | | |
| | | Total | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

S- = Initially seronegative subjects (antibody concentration below assay cut-off for anti-PT, anti-FHA, anti-PRN)

S+ = Initially seropositive (antibody concentration above assay cut-off for anti-PT, anti-FHA, anti-PRN)

Total = subjects either seropositive or ser1gative at pre-vaccination

Vaccine response to PT, FHA and PRN antigens is defined as:

For subjects with pre-vaccination antibody concentration below the assay cut-off, post-vaccination antibody concentration equal or above the assay cut-off,

For subjects with pre-vaccination antibody concentration equal or above the assay cut-off, post-vaccination antibody concentration equal or above the pre-vaccination antibody concentration

N = number of subjects with pre- and post-vaccination results available

n(%) = number(percentage) of subjects with booster response

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

\*Pre-Pri = blood sample to be collected before the first dose of the primary vaccination course

Note: The assay cut-off is 2.693 IU/mL for anti-PT, 2.046 IU/mL for anti-FHA, and 2.187 IU/mL for anti-PRN.

Template 14 Reverse cumulative curve for anti-diphtheria antibody concentration before first dose and 1 month post last dose of the primary vaccination course (ATP cohort for immunogenicity)



dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Pre-Pri = blood sample to be collected before the first dose of the primary vaccination course Post-Pri = blood sample to be collected 1 month after the last dose of the primary vaccination course Note: The groups shown in figure are indicative only. Actual groups may differ.

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 15 Number and percentage of subjects who received study vaccine doses by vaccination group (Total vaccinated cohort)

| | d | ITpa group N = | С | ontrol group N = |
|--------------------------------|---|----------------|---|------------------|
| Total number of doses received | n | % | n | % |
| 0 | | | | |
| 1 | | | | |
| 2 | | | | |
| 3 | | | | |
| Any | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

N = number of subjects in each group or in total included in the considered cohort

n(%) = number(percentage) of subjects receiving the specified total number of doses

Any = number and percentage of subjects receiving at least 1 dose

### Template 16 Compliance in returning symptom sheets (Total vaccinated cohort)

| Dose | Group | Number of doses | Doses NOT according to protocol | Number of general SS | Compliance % general SS | Number of local SS | Compliance % local SS |
|---|---|---|---|---|---|---|---|
| 1 | dTpa group | | | | | | |
| | Control group | | | | | | |
| 2 | dTpa group | | | | | | |
| | Control group | | | | | | |
| 3 | dTpa group | | | | | | |
| | Control group | | | | | | |
| Total | dTpa group | | | | | | |
| | Control group | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

SS = Symptom sheets used for the collection of local and general solicited AEs

Compliance % = (number of doses with symptom sheet return / number of administered doses) X 100

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 17 Percentage and nature of <grade 3>symptoms (solicited and unsolicited) reported during the 4-day (Days 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | Any symptom | | | ( | Genera | ıl sym | ptom | S | Local symptoms | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95% | 6 CI | | | | 95% | CI |
| | Group | N | n | % | LL | UL | N | n | % | LL | UL | N | n | % | LL | UL |
| Dose 1 | dTpa group | | | | | | | | | | | | | | | |
| | Control group | | | | | | | | | | | | | | | |
| | dTpa group | | | | | | | | | | | | | | | |
| | Control group | | | | | | | | | | | | | | | |
| Dose 3 | dTpa group | | | | | | | | | | | | | | | |
| | Control group | | | | | | | | | | | | | | | |
| Overall/dose | dTpa group | | | | | | | | | | | | | | | |
| | Control group | | | | | | | | | | | | | | | |
| Overall/subject | | | | | | | | | | | | | | | | |
| | Control group | | | | | | | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

For each dose and overall/subject:

N= number of subjects with at least 1 administered dose

n(%) = number(percentage) of subjects presenting at least 1 type of symptom whatever the study vaccine administered For overall/dose:

N= number of administered doses

n(%) = number(percentage) of doses followed by at least 1 type of symptom whatever the study vaccine administered 95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## Template 18 Percentage of solicited local symptoms reported during the 4-day (Day 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | | | | | eac | h gro | oup | ) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | dTp | a gro | up | | C | ont | rol gr | |
| | | | | | 95 | 5 % CI | | | | 9 | 5 % CI |
| Symptom | Product | Туре | N | n % | LL | UL | N | n | % | LL | UL |
| | | | Each | dose | | | | | | | |
| Pain | Total | All | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | |
| | | Grade 3 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | |
| | | Grade 2 or3 | | | | | | | | | |
| | | Grade 3 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | |
| | | Grade 3 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| Redness | Total | All | | | | | | | | | |
| (mm) | | > 5.0 | | | | | | | | | |
| ` ' | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | |
| | | > 5.0 | | | | | | | | | |
| Prevenar | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | |
| | | > 5.0 | | | | | | | | | |
| | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| Swelling | Total | All | | | | | | | | | |
| (mm) | | > 5.0 | | | | | | | | | |
| | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | |
| | | > 5.0 | | | | | | | | | |
| | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | |
| | | > 5.0 | | | | | | | | | |
| | | > 20.0 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | · | Overall/Do | ose | | • | | | | | | |
| Pain | Total | All | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | |
| | | Grade 3 | | | | | | | | | |
| | | Medical advice | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | Ì | | |
| | | Grade 2 or 3 | | | | | | | Ì | | |
| | | Grade 3 | | | | | | | İ | | |
| | | Medical advice | | | | | | | | | |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

| | | | | | | | eac | | | | | n Fin |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | ·Tns | grou | | y y | | | ol gro | un |
| | | | | | ı ı pc | | % CI | | | Onti | | % CI |
| Symptom | Product | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| oyinptoin . | Prevenar 13 | All | 11 | " | /0 | | OL | 14 | " | /0 | | OL |
| | Flevellal 13 | Grade 2 or 3 | | | | | | | | | | |
| | | Grade 3 | | | | | | | | | | |
| | | Medical advice | | | | | | - | | | - | |
| Dadaaa (mm) | Total | All | | | | | | - | | | - | |
| Redness (mm) | Total | > 5.0 | | | | | | - | | | | |
| | | > 20.0 | | | | | | - | | | | |
| | | Medical advice | | | | | | - | | | | |
| | la fa a sir da a ca | | | | | | | - | | | | |
| | Infanrix hexa | All | | | | | | | | | | |
| | | > 5.0<br>> 20.0 | | | | | | - | | | | |
| | D 40 | Medical advice | | | | | | | | | | |
| | Prevenar 13 | All | | | | | | - | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| Swelling (mm) | Total | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | | Overall/Sub | ject | | | | | | | | | |
| Pain | Total | All | | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | | |
| | | Grade 3 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | | |
| | | Grade 3 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | | |
| | | Grade 2 or 3 | | | | | | | | | | |
| | | Grade 3 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| Redness (mm) | Total | All | | | | | İ | | | | | |
| , , | | > 5.0 | | | | | 1 | | | | | |
| | | > 20.0 | | | | | | 1 | | | 1 | |
| | | Medical advice | | T | | | | 1 | T | t | | |
| | Infanrix hexa | All | | $I^-$ | | | | T | $I^-$ | | | |
| | | > 5.0 | | T | | | 1 | 1 | T | | 1 | 1 |
| | | > 20.0 | | | | | | 1 | | | <del> </del> | 1 |
| | | | | | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

| | | | Statistical Analysis Fian Fil | | | | | | | | | all I IIIc |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | eac | h gr | | | | |
| | | | | ( | dTp | a grou | лb | | C | onti | ol gr | oup |
| | | | 95 % CI | | | | | | 9 | 5 % CI | | |
| Symptom | Product | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | Prevenar 13 | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| Swelling (mm) | Total | All | | | | | | | | | | |
| | > 5.0 | | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Infanrix hexa | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |
| | Prevenar 13 | All | | | | | | | | | | |
| | | > 5.0 | | | | | | | | | | |
| | | > 20.0 | | | | | | | | | | |
| | | Medical advice | | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

For each dose and overall/subject:

N= number of subjects with at least 1 documented dose

n(%) = number(percentage) of subjects reporting the symptom at least once

For Overall/dose:

N= number of documented doses

n(%) = number(percentage) of doses followed by at least 1 type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

## Template 19 Percentage of solicited general symptoms reported during the 4-day (Days 0-3) post-vaccination period following each dose and overall (Total vaccinated cohort)

| | | | dTp | a gro | | | | Cor | ntrol gr | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 9 | % CI | | | | 95 | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | LL | UL |
| | 1 | Each | dose | 1 | | | | 1 | 1 | | |
| Drowsiness | All | | | | | | | | | | |
| | Grade 2 or 3 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| rritability | All | | | | | | | | | | |
| | Grade 2 or 3 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| oss of appetite | All | | | | | | | | | | |
| | Grade 2 or 3 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | |
| | Related | | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| Temperature/(Axillary) (°C) | All | | | | | | | | | | |
| · | >37.5 | | | | | | | | | | |
| | >38.0 | | | | | | | | | | |
| | >38.5 | | | | | | | | | | |
| | >39.0 | | | | | | | | | | |
| | >39.5 | | | | | | | | | | 1 |
| | Related | | | | | | | | | | |
| | >39*Related | | | | | | | | | | |
| | Medical advice | | | | | | | | | | |
| | Wicaldal advice | Overs | ıll/dose | | | | | | | | 1 |
| Drowsiness | All | Overe | 111/4030 | | | | | | | | 1 |
| JIOWSII1633 | Grade 2 or 3 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | 1 |
| | Related | | | | | | | | | | 1 |
| | Grade 3*Related | | | | | | | | | | 1 |
| | Medical advice | | | | | | | | | | |
| rritability | All | | | | | | | | | | - |
| rritability | Grade 2 or 3 | | | | | | | | | | 1 |
| | Grade 3 | | | | | | | | | | |
| | | | | | | | | | | | - |
| | Related | | | | | | | | | | - |
| | Grade 3*Related | | | | | | | | | | - |
| | Medical advice | | | | | | | | | | <del> </del> |
| oss of appetite | All | | | | | | | | | | <u> </u> |
| | Grade 2 or 3 | | | | | | | | | | |
| | Grade 3 | | | | | | | | | | 1 |
| | Related | | | | | | | | | | <u> </u> |
| | Grade 3*Related | | | | | | | | | | <u> </u> |
| | Medical advice | | | 1 | | | | | | l | 1 |

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

| | | | dTn | a gro | un | | olalist | | naiysis<br>i <b>trol gr</b> | 1 1 11 10 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | 4.6 | u g. o | | % CI | | | iti Oi gi | % CI |
| Symptom | Туре | N | n | % | LL | UL | N | n | % | UL |
| Temperature/(Axillary) (°C) | All | | - " | 70 | | 0_ | | -"- | /0 | <br><del>-</del> |
| Tomperature/(rixillary) ( O) | >37.5 | | | | | | | | | - |
| | >38.0 | | | | | | | | | + |
| | >38.5 | | | | | | | | | - |
| | >39.0 | | | | | | | | | 1 |
| | >39.5 | | | | | | | | | 1 |
| | Related | | | | | | | | | + |
| | >39*Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| | | Overall | /subie | ct | 1 | | | l | 1 | .1 |
| Drowsiness | All | | | | | | | | | |
| 210110111000 | Grade 2 or 3 | | | | | | | | | |
| | Grade 3 | | | | | | | | | |
| | Related | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | † |
| | Medical advice | | | | | | | | | 1 |
| Irritability | All | | | | | | | | | - |
| | Grade 2 or 3 | | | | | | | | | - |
| | Grade 3 | | | | | | | | | |
| | Related | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| Loss of appetite | All | | | | | | | | | |
| | Grade 2 or 3 | | | | | | | | | |
| | Grade 3 | | | | | | | | | |
| | Related | | | | | | | | | |
| | Grade 3*Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |
| Temperature/(Axillary) (°C) | All | | | | | | | | | |
| | >37.5 | | | | | | | | | |
| | >38.0 | | | | | | | | | |
| | >38.5 | | | | | | | | | |
| | >39.0 | | | | | | | | | |
| | >39.5 | | | | | | | | | |
| | Related | | | | | | | | | |
| | >39*Related | | | | | | | | | |
| | Medical advice | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

N= number of subjects with at least 1 documented dose

n(%) = number(percentage) of subjects reporting the symptom at least once For Overall/dose:

N= number of documented doses

n(%) = number(percentage) of doses followed by at least 1 type of symptom

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Related: Symptoms which is assessed by the investigator as related to vaccination

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

# Template 20 Percentage of Unsolicited symptoms experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) after any dose (Total vaccinated cohort)

| | | dT | pa Gro<br>N = | up | Conti | rol Gr | oup N = |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| At least 1 symptom | | | | | | | |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

At least 1 symptom = at least 1 symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n(%) = number(percentage) of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Template 21 Number (%) of subjects with serious adverse events from the Day 0 to end of the study (Total Vaccinated cohort)

| Type of Event | Primary System Organ<br>Class | Preferred Term<br>(CODE) | dΤ | pa Gr<br>N = | - | Control Group N = | | |
|---|---|---|---|---|---|---|---|---|
| | | | n* | n | % | n* | n | % |
| SAE | At least 1 symptom | | | | | | | |
| | <each soc=""></each> | <each pt=""></each> | | | | | | |
| Related SAE | At least 1 symptom | | | | | | | |
| | <each soc=""></each> | <each pt=""></each> | | | | | | |
| Fatal SAE | At least 1 symptom | | | | | | | |
| | <each soc=""></each> | <each pt=""></each> | | | | | | |
| Related Fatal SAE | At least 1 symptom | | | | | | | |
| | <each soc=""></each> | <each pt=""></each> | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

Template 22 Solicited and unsolicited adverse events experienced by subjects classified by MedDRA Primary System Organ Class and Preferred Term within the 31-day (Days 0-30) post-vaccination period - SAE excluded (Total vaccinated cohort)

| | | dT | pa Grou<br>N = | р | Control Group N= | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ<br>Class (CODE)<br>At least 1 symptom | Preferred Term (CODE) | n* | n | % | n* | n | % |
| <each soc=""></each> | <each pt="" term=""></each> | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

At least 1 symptom = at least 1 symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects with the administered dose

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

# Template 23 Number and percentage of subjects taking a concomitant medication and antipyretic medication during the 4-day (Days 0-3) follow-up period post-vaccination by dose and overall (Total vaccinated cohort)

| | | ( | dTpa gro | up | | | ( | ontrol g | roup | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 5% CI | | | | 95 | % CI |
| | N | n | % | LL | UL | N | n | % | LL | UL |
| | 1 | | Each d | ose | ' | | • | | | |
| Any | | | | | | | | | | |
| Any antipyretic | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | |
| | " | | Overall/o | dose | ' | | • | | | |
| Any | | | | | | | | | | |
| Any antipyretic | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | |
| | " | ( | Overall/su | ubject | ' | | • | | | |
| Any | | | | | | | | | | |
| Any antipyretic | | | | | | | | | | |
| Prophylactic antipyretic | | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

For each dose and overall/subject:

N= number of subjects with at least 1 administered dose

n(%) = number(percentage) of subjects who started to take the specified concomitant medication at least once during the menti1d period

For overall/dose:

N= number of administered doses

n(%) = number(percentage) of doses after which the specified concomitant medication was started at least once during the menti1d period

95% CI = exact 95% confidence interval, LL = Lower Limit, UL = Upper Limit

### Template 24 Minimum and maximum activity dates (Total vaccinated cohort)

| Visit | Minimum date | Maximum date |
|-------|--------------|--------------|
| 1 | 19JUN2007 | 29DEC2007 |
| 2 | 24JUL2007 | 08FEB2008 |
| 3 | 24AUG2007 | 18MAR2008 |
| 4 | 25MAR2008 | 22NOV2008 |

Database Lock Date = 31MAR2009

201330 [DTPA (BOOSTRIX)-048 PRI] Statistical Analysis Plan Final

### Template 25 Number of enrolled subjects by age category at visit1

| | | dTpa group<br>N = | Control group<br>N = | Total<br>N = |
|---|---|---|---|---|
| Characteristics | Categories | n | n | n |
| Age category | Infants (6 weeks – 14 weeks and 6 days) | | | |
| | Missing | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

N = Number of enrolled subjects

n = number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = subjects who are enrolled in the study but not vaccinated and for which age is unknown

### Template 26 Listing of SAEs from Day 0 up study (Total vaccinated cohort)

| Group | | | | | Verbati | Preferre | Syste | ME | Dos | Day | Duratio | Intensit | Causalit | Outcom |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | e Id | onset | X | m | d term | m | _ | - | of | n | У | У | е |
| | No. | | (Week | | | | Organ<br>Class | type | | onse | | | | |
| | | | , | | | | Olass | | | t | | | | |
| dTpa | | | | | | | | | | | | | | |
| group | | | | | | | | | | | | | | |
| Contro | | | | | | | | | | | | | | |
| I group | | | | | | | | | | | | | | |

dTpa Group = This group will consist of infants born to mothers belonging to the dTpa Group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule.

Control Group: This group will consist of infants born to mothers belonging to the Control group in study 116945 [DTPA (BOOSTRIX)-047]. All subjects in this group will receive *Infanrix hexa* co-administered with *Prevenar 13* according to the routine national immunisation schedule. For each dose and overall/subject:

Med type = Type of medical advice; HO= Hospitalisation, ER = Emergency room

### Template 27 Listing of dropouts due to AEs, SAEs and solicited symptoms (Total vaccinated cohort)

| Group | Sub. No. | Country | Gender | AE Description | SAE | Causality | Outcome | Type of discontinuation |
|---|---|---|---|---|---|---|---|---|
| dTpa<br>group | PP | Germany | F | SUBJECT DIED | Y | | Fatal | Study at visit/contact: VISIT11 (Y5) |
| Control<br>group | PP | Germany | F | SUBJECT DIED | Y | | Fatal | Study at visit/contact: VISIT11 (Y5) |